CLINICAL TRIAL: NCT01700946
Title: A Phase II Study of Therapy for Pediatric Relapsed or Refractory Precursor B-Cell Acute Lymphoblastic Leukemia and Lymphoma
Brief Title: Therapy for Pediatric Relapsed or Refractory Precursor B-Cell Acute Lymphoblastic Leukemia and Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Cookies for Kids' Cancer (Other); Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLR18; NCI-2012-00587 (Registry Identifier: NCi Clinical Trial Registration Program)
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Recurrent B-Cell Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood B-Lymphoblastic Lymphoma
Keywords: leukemia; lymphoma; Non-Hodgkins
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Dexamethasone; Vincristine; Rituximab; Clofarabine; Cyclophosphamide; Etoposide; aldesleukin; Interleukin-2; pegaspargase; Methotrexate; Mercaptopurine; Cytarabine; Mitoxantrone; Teniposide; Vinblastine; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard Risk (Active Comparator): Interventions: dexamethasone, vincristine sulfate, rituximab, clofarabine, cyclophosphamide, etoposide, aldesleukin, pegaspargase, methotrexate, mercaptopurine, cytarabine, mitoxantrone, teniposide, vinblastine, natural killer cell infusion, laboratory biomarker analysis, therapeutic hydrocortisone
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: dexamethasone; Drug: vincristine sulfate; Biological: rituximab; Drug: clofarabine; Drug: cyclophosphamide; Drug: etoposide; Biological: aldesleukin; Drug: pegaspargase; Drug: methotrexate; Drug: mercaptopurine; Drug: cytarabine; Drug: mitoxantrone; Drug: teniposide; Drug: vinblastine; Biological: natural killer cell infusion; Other: laboratory biomarker analysis; Drug: therapeutic hydrocortisone; Device: CliniMACS
- High Risk (Active Comparator): Interventions: dexamethasone, vincristine, rituximab, clofarabine, cyclophosphamide, etoposide, aldesleukin, pegaspargase, methotrexate, mercaptopurine, cytarabine, mitoxantrone, natural killer cell infusion, allogeneic hematopoietic stem cell transplantation, laboratory biomarker analysis, therapeutic hydrocortisone
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: dexamethasone; Drug: vincristine sulfate; Biological: rituximab; Drug: clofarabine; Drug: cyclophosphamide; Drug: etoposide; Biological: aldesleukin; Drug: pegaspargase; Drug: methotrexate; Drug: mercaptopurine; Drug: cytarabine; Drug: mitoxantrone; Biological: natural killer cell infusion; Other: laboratory biomarker analysis; Drug: therapeutic hydrocortisone; Procedure: allogeneic hematopoietic stem cell transplantation; Device: CliniMACS

INTERVENTIONS:
Drug: dexamethasone — given intravenously or orally
  Other Names: Decadron(R)
Drug: vincristine sulfate — given intravenously
  Other Names: Oncovin(R)
Biological: rituximab — given intravenously
  Other Names: Rituxan(R)
Drug: clofarabine — given intravenously
  Other Names: Clolar(TM); clofarex
Drug: cyclophosphamide — given intravenously
  Other Names: Cytoxan(R)
Drug: etoposide — given intravenously
  Other Names: VP-16; Vepesid(R)
Biological: aldesleukin — given subcutaneously
  Other Names: IL-2; interleukin-2; Proleukin (R)
Drug: pegaspargase — given intravenously
  Other Names: PEG-ASP; Peg-L-asparaginase; PEG-asparaginase; Oncaspar(R)
Drug: methotrexate — given intrathecally or intravenously
  Other Names: MTX; HDMTX
Drug: mercaptopurine — given orally
  Other Names: 6-MP; Purinethol(R)
Drug: cytarabine — given intrathecally or intravenously
  Other Names: Ara-C; Cytosar-U(R)
Drug: mitoxantrone — given intravenously
  Other Names: Novantrone(R)
Drug: teniposide — given intravenously
  Other Names: VM-26; Vumon(R)
  Arms: Standard Risk
Drug: vinblastine — given intravenously
  Other Names: Velban(R)
  Arms: Standard Risk
Biological: natural killer cell infusion — undergo allogeneic natural killer cell infusion
  Other Names: NK cell infusion
Other: laboratory biomarker analysis — correlative studies
Drug: therapeutic hydrocortisone — given intrathecally
  Other Names: Cortef
Procedure: allogeneic hematopoietic stem cell transplantation — undergo allogeneic HSCT
  Other Names: HSCT
  Arms: High Risk
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System

SUMMARY:
The overall objective of this protocol is to improve the cure rate of relapsed precursor B-cell acute lymphoblastic leukemia (ALL) and lymphoblastic lymphoma.

This phase II trial is studying risk-directed therapy for B-lymphoblastic leukemia or lymphoma in first relapse. Standard risk (SR) and high risk (HR) participants will receive different therapy. Treatment will consist of chemotherapy for SR participants, and chemotherapy followed by hematopoietic stem cell transplant (HSCT) for HR in first relapse. Induction therapy consists of three blocks of chemotherapy. The first block is a novel immunotherapy regimen that includes chemotherapy, rituximab and infusion of haploidentical natural killer (NK) cells. SR participants will continue to receive chemotherapy for a total duration of approximately 2 years. HR participants will be candidates for HSCT and will proceed to transplant once a suitable donor is found and their minimal residual disease (MRD) is negative.

DETAILED DESCRIPTION:
Primary objective

* To estimate the 3-year survival rate of participants with first relapse or primary refractory precursor B-cell ALL and lymphoblastic lymphoma treated with risk-directed therapy.

Secondary objectives

* To determine minimal residual disease (MRD) levels at the end of remission induction therapy for participants with relapsed precursor B-cell ALL and compare the results with those in protocol ALLR17
* To estimate levels of CD20 expression at baseline, during treatment with dexamethasone-containing chemotherapy and following rituximab treatment in Block 1 of remission induction therapy for relapsed precursor B-cell ALL.

STUDY DESCRIPTION:

The general treatment plan will consist of chemotherapy for standard-risk participants and chemotherapy followed by HSCT for high risk participants in first relapse of B-precursor ALL or lymphoblastic lymphoma. Remission induction for all participants consists of three blocks of therapy, wherein the first block is a novel immunotherapy regimen that includes cytotoxic chemotherapy, rituximab and infusion of haploidentical natural killer (NK) cells. Standard-risk patients will continue to receive chemotherapy for a total duration of approximately 2 years. High-risk patients will be candidates for HSCT and will proceed to transplant once a suitable donor is found and the patient achieves negative MRD.

Participants will be assigned to the standard arm if they experience late relapse (> or = 6 months after completion of frontline therapy) AND maximum residual disease (MRD) is <0.01% at the end of Block II of remission induction therapy. Provisional standard risk participants (i.e., late relapse) will be re-assigned to high risk if MRD is > or = 0.01% at the end of Block II. Participants with lymphoma must be in complete remission at the end of Block III.

High risk participants will meet one of the following criteria:

* Early relapse (on therapy or <6 months after completion of frontline therapy), OR
* Any relapse after hematopoietic stem cell transplant, OR
* MRD > or = 0.01% at the end of Block II of remission induction therapy, OR
* Re-emergence of MRD at any time after attaining negative MRD on this clinical trial.

Natural killer (NK) cell collection: Donors who meet eligibility criteria will undergo apheresis once. The cells obtained will be purified for CD56+ cells utilizing the CliniMACS selection system. The NK cell product will undergo quality control testing following standard operating procedures of the St. Jude Human Applications Laboratory.

OUTLINE (STANDARD RISK):

REMISSION INDUCTION:

BLOCK I: Patients receive dexamethasone orally (PO) or intravenously (IV) thrice daily (TID) on days 1-8 and 21-28; vincristine sulfate IV on days 1, 21, 28, and 35; rituximab IV on days 4, 13, 20, and 27; clofarabine, cyclophosphamide, and etoposide IV on days 6-10; aldesleukin subcutaneously (SC) once every other day (QOD) on days 11-19; and pegaspargase IV on days 21 and 35. Patients also undergo natural killer (NK) cell infusion on day 12. Patients may receive triple intrathecal therapy comprising methotrexate, therapeutic hydrocortisone, and cytarabine on days 1, 5, 8, 11, 21, and 28. Patients continue on to Block II after count recovery.

BLOCK II: Patients receive methotrexate IV over 24 hours on days 1 and 8 and mercaptopurine PO on days 1-21. Patients also receive triple intrathecal therapy on day 1. High-risk patients with negative MRD continue on to transplantation. All patients with positive MRD continue on to Block III after count recovery.

BLOCK III: Patients receive cytarabine IV over 2 hours twice daily (BID) on days 1-4 and mitoxantrone hydrochloride IV over 1 hour on days 3-5. Patients also receive triple intrathecal therapy on day 7.

INTERIM CONTINUATION (for patients unable to tolerate dose intensive chemotherapy): Patients receive etoposide and cyclophosphamide IV on day 1, methotrexate IV on day 8, mercaptopurine PO on days 8-14, teniposide and cytarabine IV on day 15, dexamethasone PO TID on days 22-26, and vinblastine IV on day 22.

RE-INDUCTION THERAPY: Patients receive clofarabine, cyclophosphamide, and etoposide IV on days 1-5; dexamethasone PO on days 1-6; and pegaspargase on days 6 and 20 and vincristine sulfate IV on days 6, 13, and 20. Patients may also receive triple intrathecal therapy on days 1 and 15. Patients continue on to continuation treatment after count recovery.

CONTINUATION TREATMENT: Patients receive methotrexate IV over 2 hours on day 1 and mercaptopurine PO on days 1-7 of weeks 1, 2, 5, and 6; teniposide and cytarabine IV on day 1 of weeks 3 and 7; vincristine sulfate IV on day 1 of week 4; dexamethasone PO TID on days 1-5 of weeks 4 and 8; and vinblastine IV on day 1 of week 8. Treatment repeats every 8 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity. Patients may also receive triple intrathecal therapy on day 1 of week 1 of all courses and day 1 of week 5, courses 1-5.

Due to the unavailability of the drug Teniposide (VM-26), etoposide (VP-16) will be substituted for the remaining doses for patients currently on this study. The protocol Section 5.1.3 allows this substitution.

OUTLINE: GROUP 2 (high risk defined as participants not meeting the standard risk criteria noted above):

Patients receive Remission Induction (Blocks I, II, and III) treatment as described above for Group 1. Patients then undergo allogeneic hematopoietic stem cell transplantation (HSCT) as soon as they have negative MRD. Patients with negative MRD may continue chemotherapy until a suitable donor is found.

After completion of study treatment, patients are followed up every 4 months for 1 year, every 6 months for 1 year, and then yearly for up to 10 years.

ELIGIBILITY:
INCLUSION CRITERIA:

* Must have relapsed or refractory precursor B-cell acute lymphoblastic leukemia or acute lymphoblastic lymphoma.
* Participants with leukemia must meet one of the following:

  1. In first hematologic relapse, defined as the reappearance (in a patient who has previously achieved remission) of leukemia blasts in the bone marrow or peripheral blood, OR
  2. Refractory to one or two courses of frontline induction therapy (≥ 5% blasts in the bone marrow or peripheral blood confirmed by flow cytometric analysis).
* Participant with lymphoma must meet one of the following:

  1. In first relapse, OR
  2. Refractory to one or two courses of frontline induction therapy with measurable disease

     * Should flow cytometric analyses suggest relapse (by the reappearance of a similar immunophenotype to the original leukemia) in the presence of <5% blasts morphologically, a repeat bone marrow test is recommended to confirm relapse.
     * Molecular or genetic relapse is characterized by the reappearance of a cytogenetic or molecular abnormality.
     * Early relapse is defined as relapse on therapy or < 6 months after completion of frontline therapy. Late relapse is defined as relapse occurring ≥ 6 months after completion of frontline therapy.
* Participant's age is < 22 years at time of enrollment (e.g. participant is eligible until 22nd birthday).
* Prior therapy:

  1. There is no waiting period for participants who relapse while receiving frontline therapy and are free from side effects attributable to such therapy.
  2. Emergent radiation therapy, one dose of intrathecal chemotherapy, and up to 7 days of steroids for treatment of relapse are permitted before start of treatment in participants who relapse after completion of frontline therapy.
  3. At least 90 days have elapsed since bone marrow transplant and participant is off immune suppression for a minimum of 2 weeks, if applicable. Participants with ALL or NHL who were transplanted in first remission are eligible for this study.

Organ function requirements

* Hepatic: Total bilirubin ≤ upper limit of normal (ULN) for age, or if total bilirubin is > ULN, direct bilirubin ≤ 1.4 mg/dl
* Cardiac: Shortening fraction ≥ 28%
* Renal: Glomerular filtration rate >50cc/min/1.73 m^2, OR maximum serum creatinine (SC) based on age as follows:

  * If age is 1 to 2 years, then maximum SC is 0.6 mg/dL
  * If age is 2 to 6 years, then maximum SC is 0.8 mg/dL
  * If age is 6 to 10 years, then maximum SC is 1 mg/dL
  * If age is 10 to <13 years, then maximum SC is 1.2 mg/dL
  * If age is 13 to 16 years, then maximum SC is 1.5 mg/dL for males and 1.4 mg/dL for females
  * If age is >16 years, then maximum SC is 1.7 mg/dL for males and 1.4 mg/dL for females

EXCLUSION CRITERIA:

* Leukemia participants ages 1 to 5 years with induction failure AND favorable cytogenetics (i.e., hyperdiploidy defined as DNA index ≥1.16 or modal chromosome number ≥51, or ETV6-RUNXI).
* Hepatitis B or HIV infection.
* Pregnant or breast-feeding
* Inability or unwillingness or research participant or legal guardian/representative to give written informed consent.

INCLUSION CRITERIA FOR NK CELL DONORS:

* Donor is at least 18 years of age.
* Donor is a family member.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04-15 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Rady Children's Hospital and Health Center, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty (80) participants were enrolled on study. Forty-two (42) participants for the outcome measures and thirty-eight (38) donors who are not included in the analysis.
Groups:
- STANDARD RISK: 1. Late relapse (≥ 6 months after completion of frontline therapy) AND
  2. MRD < 0.01% at the end of Block II of remission induction therapy.
  Provisional standard risk participants (i.e., late relapse) will be re-assigned to High risk if MRD ≥ 0.01% at the end of Block II.
  Participants with lymphoma must be in complete remission at the end of Block III.
- HIGH RISK: 1. Early relapse (on therapy or < 6 months after completion of frontline therapy), OR
  2. Any relapse after hematopoietic stem cell transplant, OR
  3. MRD ≥ 0.01% at the end of Block II of remission induction therapy, OR
  4. Re-emergence of MRD at any time after attaining negative MRD on ALLR18
Period: Overall Study
Arm/Group | STANDARD RISK | HIGH RISK
Started | 18 | 24
Completed | 7 | 7
Not Completed | 11 | 17
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 7 | 12
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Failed to achieve Complete Remission after Induction Block III | 0 | 2
Not completed — Relapse | 2 | 1
Not completed — Unacceptable toxicity | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled on study.
Groups:
- Total: Total of all reporting groups
Arm/Group | STANDARD RISK | HIGH RISK | Total
Number analyzed (Participants) | 18 | 24 | 42
Age, Customized [Count of Participants; unit: Participants]
  1 to 9 years | 6 | 16 | 22
  >=10 years | 12 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 11 | 19 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2 | 3 | 5
  White | 13 | 17 | 30
  Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: 3-year Overall Survival Rate of Patients With Relapsed ALL
Description: Estimate the 3-year survival rate of participants with first relapse or primary refractory precursor B-cell ALL treated with risk-directed therapy.
Time Frame: 3 years of follow-up since the on-study date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Patients Enrolled on the Study: All patients who received the protocol-specified therapy.
Arm/Group | STANDARD RISK | HIGH RISK | All Patients Enrolled on the Study
Number analyzed (Participants) | 18 | 24 | 42
percentage of participants | 94.4 [66.6 to 99.2] | 55.5 [33.0 to 73.2] | 72.63 [55.95 to 83.85]
Statistical Analysis 1: Comparison: STANDARD RISK vs HIGH RISK; Test type: Superiority; p = 0.035, Log Rank

2. Primary Outcome: 3-year Event-free Survival Rates in Patients With Relapsed ALL
Description: Estimate the 3-year event-free survival rate of participants with first relapse or primary refractory precursor B-cell ALL treated with risk-directed therapy.
Time Frame: 3 years of follow-up since the on-study date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | STANDARD RISK | HIGH RISK | All Patients Enrolled on the Study
Number analyzed (Participants) | 18 | 24 | 42
percentage of participants | 83.3 [56.8 to 94.3] | 55.7 [33.2 to 73.4] | 67.83 [51.04 to 79.9]
Statistical Analysis 1: Comparison: STANDARD RISK vs HIGH RISK; Test type: Superiority; p = 0.105, Log Rank

3. Secondary Outcome: Proportion of Participants With Positive Minimal Residual Disease
Description: To determine minimal residual disease (MRD) levels at the end of remission induction therapy for participants with relapsed precursor B-cell ALL and compare the results with those in protocol ALLR17 (NCT00186875).
Time Frame: At end of induction (approximately 3 months)
Population: On ALLR18, a total of 42 patients enrolled. Of them, 24 patients had MRD data at the end of Remission Induction. On ALLR17, a total of 40 patients enrolled. Of them, 32 patients had MRD data at the end of Remission Induction
Measure: Count of Participants; unit: Participants
Groups:
- ALLR18; ALLR17: All patients who had MRD data at the end of Remission Induction
Arm/Group | STANDARD RISK | HIGH RISK | ALLR18 | ALLR17
Number analyzed (Participants) | 14 | 10 | 24 | 32
Participants
  MRD end-induction: Negative | 14 | 6 | 20 | 22
  MRD end-induction: Positive | 0 | 4 | 4 | 10
Statistical Analysis 1: Comparison: ALLR18 vs ALLR17; Test type: Superiority; p = 0.1181, Fisher Exact

4. Secondary Outcome: Mean of CD20 Expression Levels
Description: To estimate mean levels of CD20 expression at baseline, during treatment with dexamethasone-containing chemotherapy and following rituximab treatment in Block I of remission induction therapy for relapsed precursor B-cell ALL.
Time Frame: Baseline and at the end of Block I (approximately 5 weeks after the on-study date)
Population: Of the 42 patients enrolled, 34 patients had At Baseline data; 42 patients had data At Block I
Measure: Mean (Standard Error); unit: percentage of CD20 Antigen
Arm/Group | STANDARD RISK | HIGH RISK | All Patients Enrolled on the Study
Number analyzed (Participants) | 18 | 24 | 42
percentage of CD20 Antigen
  At Baseline: number analyzed (Participants) | 14 | 20 | 34
  At Baseline | 31.10 (9.82) | 39.82 (7.9) | 36.23 (6.11)
  At Block I | 18.54 (4.93) | 20.10 (3.44) | 19.43 (2.85)

5. Secondary Outcome: Median CD20 Expression Levels
Description: To estimate median levels of CD20 expression at baseline, during treatment with dexamethasone-containing chemotherapy and following rituximab treatment in Block I of remission induction therapy for relapsed precursor B-cell ALL.
Time Frame: Baseline and at the end of Block I (approximately 5 weeks after the on-study date)
Population: Of the 42 patients enrolled, 34 patients had At Baseline data; 42 patients had data At Block I
Measure: Median (Inter-Quartile Range); unit: percentage of CD20 Antigen
Arm/Group | STANDARD RISK | HIGH RISK | All Patients Enrolled on the Study
Number analyzed (Participants) | 18 | 24 | 42
percentage of CD20 Antigen
  At Baseline: number analyzed (Participants) | 14 | 20 | 34
  At Baseline | 16.40 [3.30 to 36.8] | 23.13 [8.75 to 67.25] | 22.0 [4.30 to 61.20]
  At Block 1 | 11.83 [1.50 to 22.15] | 19.58 [2.6 to 30.67] | 15.58 [1.50 to 30.13]

ADVERSE EVENTS:
Time Frame: Through one month after therapy completion, approximately 22 months. If participant proceeds to transplant, until the first day of conditioning therapy.
Arm/Group | STANDARD RISK | HIGH RISK | All Patients Enrolled on the Study
All-Cause Mortality (participants affected / at risk) | 3/18 | 10/24 | 13/42
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/24 | 1/42
Other Adverse Events (participants affected / at risk) | 18/18 | 23/24 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STANDARD RISK (N=18) | HIGH RISK (N=24) | All Patients Enrolled on the Study (N=42)
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | STANDARD RISK (N=18) | HIGH RISK (N=24) | All Patients Enrolled on the Study (N=42)
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 22 | 40
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 23 | 40
Alanine aminotransferase increased (Investigations) | 18 | 21 | 39
Aspartate aminotransferase increased (Investigations) | 17 | 21 | 38
Hypokalemia (Metabolism and nutrition disorders) | 15 | 20 | 35
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 19 | 35
Hypophosphatemia (Metabolism and nutrition disorders) | 15 | 20 | 35
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 17 | 34
Nausea (Gastrointestinal disorders) | 15 | 19 | 34
Hyponatremia (Metabolism and nutrition disorders) | 15 | 18 | 33
Mucositis oral (Gastrointestinal disorders) | 14 | 14 | 28
Anorexia (Metabolism and nutrition disorders) | 12 | 13 | 25
Constipation (Gastrointestinal disorders) | 11 | 11 | 22
Hypermagnesemia (Metabolism and nutrition disorders) | 9 | 12 | 21
Infections and infestations - Other, specify (Infections and infestations) | 8 | 12 | 20
Fatigue (General disorders) | 9 | 11 | 20
Hypertension (Vascular disorders) | 7 | 12 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 14 | 19
Upper respiratory infection (Infections and infestations) | 9 | 10 | 19
Blood bilirubin increased (Investigations) | 7 | 11 | 18
Headache (Nervous system disorders) | 5 | 12 | 17
Abdominal pain (Gastrointestinal disorders) | 10 | 6 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 11 | 15
Diarrhea (Gastrointestinal disorders) | 4 | 10 | 14
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 8 | 14
Vomiting (Gastrointestinal disorders) | 5 | 9 | 14
Enterocolitis infectious (Infections and infestations) | 6 | 8 | 14
Sepsis (Infections and infestations) | 10 | 3 | 13
Neuralgia (Nervous system disorders) | 7 | 5 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 6 | 12
Skin infection (Infections and infestations) | 6 | 5 | 11
Pain (General disorders) | 5 | 5 | 10
Infusion related reaction (General disorders) | 6 | 4 | 10
Allergic reaction (Immune system disorders) | 3 | 6 | 9
Mucosal infection (Infections and infestations) | 5 | 3 | 8
Colitis (Gastrointestinal disorders) | 5 | 3 | 8
Alkaline phosphatase increased (Investigations) | 4 | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8
Fever (General disorders) | 3 | 4 | 7
Serum amylase increased (Investigations) | 4 | 3 | 7
Urinary tract infection (Infections and infestations) | 3 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Hypernatremia (Metabolism and nutrition disorders) | 1 | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 6
Lipase increased (Investigations) | 3 | 3 | 6
Hypotension (Vascular disorders) | 4 | 2 | 6
GGT increased (Investigations) | 4 | 2 | 6
Agitation (Psychiatric disorders) | 3 | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1 | 6
Rectal pain (Gastrointestinal disorders) | 1 | 4 | 5
Weight loss (Investigations) | 3 | 2 | 5
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 2 | 5
Hyperuricemia (Metabolism and nutrition disorders) | 3 | 2 | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 2 | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Chills (General disorders) | 3 | 1 | 4
Lung infection (Infections and infestations) | 4 | 0 | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 3 | 4
Blurred vision (Eye disorders) | 3 | 1 | 4
Catheter related infection (Infections and infestations) | 3 | 1 | 4
Anxiety (Psychiatric disorders) | 3 | 1 | 4
Depression (Psychiatric disorders) | 2 | 2 | 4
Acidosis (Metabolism and nutrition disorders) | 3 | 0 | 3
Eye pain (Eye disorders) | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 1 | 3
Hematoma (Vascular disorders) | 0 | 3 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 2 | 3
Non-cardiac chest pain (General disorders) | 2 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 0 | 6
Anorectal Infection (Infections and infestations) | 2 | 3 | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Meningitis (Infections and infestations) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 2
Encephalopathy (Nervous system disorders) | 2 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Dry eye (Eye disorders) | 1 | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 2
Bladder infection (Infections and infestations) | 1 | 1 | 2
Hematuria (Renal and urinary disorders) | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Encephalitis infection (Infections and infestations) | 1 | 0 | 1
Papulopustular rash (Infections and infestations) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 1
Bone infection (Infections and infestations) | 1 | 0 | 1
Infective myositis (Infections and infestations) | 1 | 0 | 1
Lip infection (Infections and infestations) | 1 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Cardiac troponin T increased (Investigations) | 1 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 2
Edema face (General disorders) | 0 | 2 | 2
Otitis media (Infections and infestations) | 0 | 2 | 2
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2 | 2
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT01700946/Prot_SAP_000.pdf